CLINICAL TRIAL: NCT06825273
Title: Clinical Evaluation of 3-D Printed Partial Denture Space Maintainer and Its Impact on Children's Oral Health Status: A Randomized Controlled Clinical Crossover Study
Brief Title: Clinical Evaluation of 3-D Printed Partial Denture Space Maintainer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Shaimaa Shaban Mohamed El-desouky, assistant professor of pediatric dentistry, Tanta University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: # R-PED-1-25-3169
Record Dates: First submitted 2025-02-08; First posted 2025-02-13 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Space Maintenance; Gingival Health
Keywords: partial denture space maintainer; 3-D printing; plaque index; gingival index

STUDY DESIGN:
Intervention Model Description: A Randomized Controlled Clinical Crossover Study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- conventional acrylic partial denture space maintainer (Active Comparator): an elastomeric impression will be done to produce a plaster cast then a conventional acrylic partial space maintainer will be fabricated and delivered for the child patient.
- 3-D printed partial denture space maintainer (Experimental): A 3-D intraoral scanner will be used to produce digital models. STL file will be used to design a 3-D printed partial denture space maintainer which will be delivered to the child patient.

INTERVENTIONS:
Other: space maintainer — 3-D printed partial denture space maintainer will designed for each child patient who has premature loss of primary teeth after doing intraoral scanning
Other: space maintainer — a conventional impression will be done for a child patient with premature loss of his primary teeth, then a plaster model will gained. A conventional acrylic partial denture will be designed and delivered to the patient.

SUMMARY:
Primary dentition is the most suitable space maintainer for permanent teeth. However, as infants often lose their primary teeth too soon, using a space maintainer is the most efficient, long-lasting, and economical way to prevent malocclusions and function impairment in the future. Regarding personalized appliances, space maintainers in digital pediatric dentistry have made significant progress. Digital technology decreases the manual manufacturing stages that take a long time and increases the reliability and durability of digital fabrication procedures.

ELIGIBILITY:
Inclusion Criteria:

* apparently, healthy cooperative children having recent premature loss of lower primary molars
* the permanent successors of the lost primary molars were not expected to erupt within 6 months
* Angle's class 1 occlusion with normal primary molar relation
* Presence of teeth on the mesial and distal side of the edentulous area
* Absence of para-functional habits or abnormal occlusion conditions such as crossbite, open bite, or deep bite.
* Radiographically, presence of permanent successors.
* parents and children were accepting the new treatment modality.

Exclusion Criteria:

* children exhibited poor oral hygiene, para-functional oral habits, severe crowding, space loss, and abnormal occlusion
* Extraction of primary molars exceeding three months.
* Radiographically, absence of permanent successor.
* uncooperative children

Ages: 7 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
clinical evaluation | three months
  the clinical performance of the partial denture space maintainers in the recall visits will be to assess: the Fracture of the space maintainer, and Lost or missing
gingival health | three months
  using a Williams periodontal probe, gingival index will be evaluated according to the following criteria:
  * 0: Healthy gingiva.
  * 1: There is mild inflammation, discoloration and edema, no bleeding on probing.
  * 2: Moderate inflammation, marked redness, edema, and bleeding on probing.
  * 3: Severe inflammation, prominent redness and edema, ulceration, spontaneous bleeding tendency.
plaque index | three months
  using a Williams periodontal probe, the plaque index will be assessed using the Silness-Loe plaque index: 0: Absence of microbial plaque, 1: Thin film of microbial plaque along the free gingival margin, 2: Moderate accumulation with plaque in the sulcus, 3: Large amount of plaque in the sulcus or pocket along the free gingiva margin.

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - pediatric dentistry department, faculty of dentistry, Tanta university, Tanta
  - Tanta University, Tanta

REFERENCES:
- [Background] Guo H, Wang Y, Zhao Y, Liu H. Computer-aided design of polyetheretherketone for application to removable pediatric space maintainers. BMC Oral Health. 2020 Jul 10;20(1):201. doi: 10.1186/s12903-020-01184-6. PMID 32650758
- [Background] Dhanotra KG, Bhatia R. Digitainers-Digital Space Maintainers: A Review. Int J Clin Pediatr Dent. 2021;14(Suppl 1):S69-S75. doi: 10.5005/jp-journals-10005-2040. PMID 35082471
- [Background] Loe H. The Gingival Index, the Plaque Index and the Retention Index Systems. J Periodontol. 1967 Nov-Dec;38(6):Suppl:610-6. doi: 10.1902/jop.1967.38.6.610. No abstract available. PMID 5237684